CLINICAL TRIAL: NCT01369082
Title: Extended Follow-Up After Islet Transplantation in Type 1 Diabetes (CIT-08)
Brief Title: Extended Follow-Up After Islet Transplantation in T1D
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Clinical Islet Transplantation Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT CIT-08
Record Dates: First submitted 2011-06-03; First posted 2011-06-08 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes (T1D); Islet Transplantation
Keywords: islet allograft function; c-peptide production; maintenance immunosuppressive medications
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Tacrolimus; Sirolimus; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants are given the option to provide consent for:
  1. the collection and storage of blood samples for future research studies
  2. the collection and storage of blood samples for future genetic (i.e., DNA) testing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CIT Islet Transplantation Recipients: Subjects who received an islet-cell transplant for Type 1 Diabetes (T1D) while enrolled in one of the Clinical Islet Transplantation (CIT) parent studies and continue to have islet graft function. All subjects will continue immunosuppressive medications under CIT08. Detailed follow-up evaluations including but not limited to islet function will occur on an annual basis.
  The immunosuppressive medications (e.g., tacrolimus, sirolimus, cyclosporine, mycophenolate mofetil [MMF], mycophenolic sodium) in this study are obtained by prescription unless provided by the study through the drug distributor. Generic brands are allowed, when available. Antibacterial, antifungal, and antiviral prophylaxis, insulin therapy, and other standard therapies will be provided per site-specific practices.
  Interventions: Drug: Maintenance Immunosuppressive Treatment

INTERVENTIONS:
Drug: Maintenance Immunosuppressive Treatment — All immunosuppressive and immunomodulatory therapies are used presently to prevent rejection of transplanted islet cells. The agents listed are those used in the parent trials and continued in this trial, CIT08.
  Other Names: tacrolimus; Prograf®; FK506; sirolimus; rapamycin; Rapamune®; cyclosporine; Neoral®; mycophenolate mofetil (MMF); CellCept®; mycophenolic sodium; Myfortic®

SUMMARY:
The purpose of this study is to provide patients who have received at least one islet transplant as a previous participant in a Clinical Islet Transplantation Consortium (CIT) clinical trial with maintenance immunosuppressive medications and to collect information about the safety of the medications and islet function.

DETAILED DESCRIPTION:
After islet-cell transplantation in the CIT studies*, each subject receives maintenance immunosuppressive medications.

The purpose of this protocol is to collect additional follow-up for safety and efficacy from CIT subjects with graft function after their completion in their CIT parent study. It is expected that most subjects will retain measurable islet function and, in the islet-alone studies, continue to receive immunosuppressive medications at the time of completing their CIT parent study.

*CIT parent studies: CIT02 (NCT00464555), CIT03 (NCT00434850), CIT04 (NCT00468403), CIT05 (NCT00468442), CIT06 (NCT00468117), and CIT07 (NCT00434811)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received an islet transplant during participation in the following Clinical Islet Transplantation (CIT) parent studies: CIT02 (NCT00464555), CIT03 (NCT00434850), CIT04 (NCT00468403), CIT05 (NCT00468442), CIT06 (NCT00468117), and CIT07 (NCT00434811)
* A functioning pancreatic islet graft (e.g., absence of graft failure as defined in parent study) requiring immunosuppression
* Willingness of participants to continue to use an approved method of contraception during and 4 months after study participation
* Ability to provide written informed consent
* Resident of the United States of America
* Documentation of the existence or lack of health insurance coverage and whether immunosuppressants are covered.

Exclusion Criteria:

* For female subjects-Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation
* For male subjects-Intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
* Received an islet transplant in a non-CIT research study
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort from Clinical Islet Transplantation (CIT) parent studies (refer to inclusion criteria) who continue:
  * to have islet graft function and
  * are on prescribed immunosuppression medications to prevent rejection of their transplant.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Duration of sustained islet allograft function | Month 36,48,60,72,84,96,108,120,132 and 144 status post last islet transplant
  A C-peptide >/= 0.3 ng/mL at 0, 60, or 90 minutes after a Mixed-Meal Tolerance Test (MMTT) will be considered evidence of insulin production by transplanted islets

SECONDARY OUTCOMES:
Serum creatinine and calculated eGFR at each annual study visit | Month 36,48,60,72,84,96,108,120,132 and 144 status post last islet transplant
  Measured as part of each annual follow-up evaluation
Incidence of serious adverse events (SAEs) during the 12-month period preceding each annual study visit | Month 36,48,60,72,84,96,108,120,132 and 144 status post last islet transplant
  Insulin usage will be estimated from the one-week self report values
Insulin requirements during a one-week period preceding each annual study visit | Month 36,48,60,72,84,96,108,120,132 and 144 status post last islet transplant
  Insulin usage will be estimated from the one-week self report values
Incidence of severe hypoglycemic events during the 12-month period preceding each annual study visit | 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months, 120 months, 132 months and 144 months
  Numbers of severe hypoglycemic events will be estimated from the self report values obtained at each follow-up visit. Defined as an event with one of the following symptoms: memory loss; confusion; uncontrollable behavior; irrational behavior; unusual difficulty in awakening; suspected seizure; seizure; loss of consciousness; or visual symptoms, in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54 mg/dL (3.0 mmol/L) or prompt recovery after oral carbohydrate, IV glucose, or glucagon administration.
HbA1c levels at each annual study visit | Month 36,48,60,72,84,96,108,120,132 and 144 status post last islet transplant
  Glycosylated hemoglobin test determination during each follow-up visit
Incidence of all-cause mortality | By month 144 status post last islet transplant
Donor-specific alloantibodies | By month 144 status post last islet transplant
  Subjects with confirmed graft failure will continue with annual study visits; however, metabolic assessments should not be completed. Subjects who were enrolled in islet-alone parent studies and who experience graft failure and subsequently stop immunosuppression will have alloantibody assessed 3 months after their last dose of immunosuppression.

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Hering, MD, Principal Investigator — University of Minnesota; Ali Naji, PhD, Principal Investigator — University of Pennsylvania; Camillo Ricordi, MD, Principal Investigator — University of Miami; Andrew Posselt, MD, PhD, Principal Investigator — University of California, San Francisco; Nicole Turgeon, MD, Principal Investigator — Emory University; Xunrong Luo, MD, PhD, Principal Investigator — Northwestern University
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Rickels MR, Liu C, Shlansky-Goldberg RD, Soleimanpour SA, Vivek K, Kamoun M, Min Z, Markmann E, Palangian M, Dalton-Bakes C, Fuller C, Chiou AJ, Barker CF, Luning Prak ET, Naji A. Improvement in beta-cell secretory capacity after human islet transplantation according to the CIT07 protocol. Diabetes. 2013 Aug;62(8):2890-7. doi: 10.2337/db12-1802. Epub 2013 Apr 29. PMID 23630300
- [Background] Shapiro AM, Ricordi C, Hering BJ, Auchincloss H, Lindblad R, Robertson RP, Secchi A, Brendel MD, Berney T, Brennan DC, Cagliero E, Alejandro R, Ryan EA, DiMercurio B, Morel P, Polonsky KS, Reems JA, Bretzel RG, Bertuzzi F, Froud T, Kandaswamy R, Sutherland DE, Eisenbarth G, Segal M, Preiksaitis J, Korbutt GS, Barton FB, Viviano L, Seyfert-Margolis V, Bluestone J, Lakey JR. International trial of the Edmonton protocol for islet transplantation. N Engl J Med. 2006 Sep 28;355(13):1318-30. doi: 10.1056/NEJMoa061267. PMID 17005949
- See also: National Institute of Allergy and Infectious Diseases — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Clinical Islet Transplantation Consortium — http://www.citisletstudy.org/